CLINICAL TRIAL: NCT06136091
Title: Mechanisms Underlying Asthma Symptoms and Exacerbations Examined Across T2 Status in Children (CHEETAH) (CAUSE-03)
Brief Title: Protocol CAUSE-03 / CHEETAH
Acronym: CHEETAH
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: DAIT CAUSE-03
Record Dates: First submitted 2023-10-16; First posted 2023-11-18 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Asthma
Keywords: Asthma; Observational study; Children
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma/serum, Peripheral blood mononuclear cells (PBMCs), urine, stool, and nasal epithelial cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthma group: Participants ages 6 to 17 year old in the asthma group will be seen in clinic quarterly for one year, during periods of disease control when they are not on systemic corticosteroids (SCS)
- Non-asthma group: Participants in the non-asthma group will be seen at two scheduled visits in clinic at 3 and 12 months and will have telephone visits at 6 and 9 months

SUMMARY:
This is a one-year longitudinal, observational study of 250 urban children and adolescents with asthma and 60 without asthma, ages 6-17 years old.

Participants with asthma will require daily controller therapy with inhaled corticosteroids ICS (at least Step 2 therapy). Those without asthma cannot have used asthma medications in the year prior to enrollment and cannot demonstrate bronchodilator reversibility at baseline. Phenotypic characteristics will be established at baseline, and the participants will be seen at scheduled visits over 12 months. Each participant will be asked to monitor and self-report cold symptoms and will be asked to complete up to three cold visits

ELIGIBILITY:
Inclusion Criteria:

1. Participant and/or parent guardian must be able to understand and provide informed consent and assent
2. Have a primary place of residence in one of the pre-selected recruitment census tracts as outlined in the Protocol CAUSE-03 Manual of Operations (MOP)

   a. Participants who do not live in the pre-selected census tracts but live within the Office of Management and Budget (OMB) defined Metropolitan Statistical Area and have publicly funded health insurance will qualify for inclusion
3. Either:

   1. Have had a diagnosis of asthma made > 1 year prior to recruitment; participants who received an asthma diagnosis by a clinician <= 1 year prior to recruitment must report that their respiratory symptoms were present for more than 1 year prior to recruitment (asthma group), or
   2. No report of ever being diagnosed with asthma (non-asthma group)
4. Either:

   1. Require at least Step 2 therapy at the Screening/Enrollment Visit (asthma group), or
   2. Have not used any asthma medications in the prior year (non-asthma group)
5. Are able to perform acceptable and repeatable spirometry per American Thoracic Society (ATS) criteria prior to enrollment
6. Have documentation of current medical insurance with prescription coverage at the Screening/Enrollment Visit
7. Participant and/or parent guardian has a smartphone compatible with the study electronic Patient Reported Outcomes (ePRO) system, Medidata Patient Cloud, and is willing to download one application for study use

Exclusion Criteria:

1. Parent or guardian is not able or willing to give written informed consent or comply with study protocol
2. Have concurrent medical problems that would require systemic corticosteroids or other immunomodulators during the study
3. Are currently receiving immunotherapy
4. Are currently receiving treatment with a biologic therapy or have received a biologic therapy within 3 months prior to enrollment
5. Are currently requiring greater than fluticasone 500 mcg bid plus Long-Acting Beta Agonists (LABA) one puff twice daily or its equivalent plus Long Acting Muscarinic Antagonists (LAMA) and/or individuals using oral corticosteroids daily or every other day for more than 14 days at the time of the Screening/Enrollment Visit
6. Are currently pregnant or lactating, or plan to become pregnant during the time of study participation. Females of child-bearing potential (post-menarche) must be abstinent or use a medically acceptable birth control method throughout the study (i.e., oral subcutaneous, mechanical, or surgical contraception)
7. Have a known, pre-existing clinically important lung condition other than asthma.
8. Have a current malignancy or previous history of cancer in remission for less than 12 months prior to enrollment
9. Have a known immunodeficiency disease
10. Use of investigational drugs within 4 weeks of enrollment
11. Have past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the site investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study
12. If in the asthma group, will not allow the study clinician, an asthma specialist, to manage their disease for the duration of the study or who are not willing to change their asthma medications to follow Protocol CAUSE-03 CHEETAH
13. If in the non-asthma group, having bronchodilator reversibility (improvement in Forced expiratory volume in 1 second (FEV1) with albuterol > = 10%) at the Screening/Enrollment visit
14. Have had a life-threatening asthma exacerbation in the last 2 years requiring intubation, mechanical ventilation or resulting in a hypoxic seizure. Potential participants may be reassessed as outlined in the Protocol CAUSE-03 Manual of Procedures (MOP)

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Approximately 250 urban children and adolescents with asthma (requiring daily controller therapy with Inhaled corticosteroid (ICS) (at least Step 2 therapy) and approximately 60 urban children and adolescents without asthma
Sampling Method: Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Asthma disease activity measured by the number of exacerbations during the 12-month observation period | Month 0 to Month 12

SECONDARY OUTCOMES:
Childhood Asthma Severity Index (CASI) | Month 0 to Month 12
  measured on a scale from 0 to 20 with smaller scores indicate a better outcome.
Modified Rhinitis Symptom Utility Index (MRSUI) | Month 0 to Month 12
  measured by assessing the frequency and severity (degree of bothering: not bothered, somewhat bothered, bothered a lot) of the participant's (1) stuffy or blocked nose, (2) runny nose, (3) sneezing, (4) itchy, watery eyes, and (5) itchy nose or throat over the preceding 14-day period
Wisconsin Upper Respiratory Symptom Survey for Kids (WURSS-K) | Month 0 to Month 12
  measured on a scale from 0 to 42 with higher scores indicating a worse outcome (high symptoms and high functional impairment)
Quality of life measured by the pediatric patient-reported (ages 8-17) or proxy-reported (ages 6-7) Patient-Reported Outcomes Measurement Information System (PROMIS) Asthma Impact Short Forms | Month 0 to Month 12
  The outcome measure is a score on a scale from 8 - 40 with higher scores indicating a worse outcome (more severe asthma symptoms).
Post-bronchodilator forced expiratory volume in 1 second (FEV1) for asthma group | Month 3 to Month 12
Post-bronchodilator forced expiratory volume in 1 second (FEV1) for non-asthma group | At Month 0
Post-bronchodilator forced vital capacity (FVC) for asthma group | Month 3 to Month 12
Post-bronchodilator forced vital capacity (FVC) for non-asthma group | At Month 0
Bronchodilator reversibility asthma group in the asthma group, measured by the percent change in FEV1 with albuterol | Month 3 to Month 12
Bronchodilator reversibility in the non-asthma group, measured by the percent change in FEV1 with albuterol | At Month 0

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Liu, M.D., Study Chair — Children's Hospital Colorado: Allergy Program; Matthew C. Altman, M.D., M.Phil., Study Chair — Benaroya Research Institute at Virginia Mason: Systems Immunology Division
Locations (8):
- United States (8):
  - Children's Hospital Colorado: Allergy Program, Aurora, Colorado
  - Children's National Medical Center: Children's Research Institute, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago: Division of Allergy and Immunology, Chicago, Illinois
  - Boston University School of Medicine: Pulmonary Center, Boston, Massachusetts
  - Boston Children's Hospital: Department of Immunology, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai: Division of Clinical Immunology, Immunology Institute, New York, New York
  - Columbia University Medical Center: Division of Pediatric Pulmonology, New York, New York
  - Cincinnati Children's Hospital Medical Center: Asthma Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: On average, within 24 months after database lock for the trial.
Access Criteria: Open access.
URL: https://www.immport.org/home

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation — https://www.niaid.nih.gov/about/dait